CLINICAL TRIAL: NCT04517500
Title: A Home-based Intervention to Promote Mindful Breathing Awareness Through Pursed-lip Breathing Training for COPD Patients
Brief Title: A Home-based Module to Promote Mindful Breathing Awareness for COPD Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); Minnesota HealthSolutions (Industry)
Responsible Party: Principal Investigator, Roberto P. Benzo, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 19-012772; 2R44AT009665-02 (NIH)
Record Dates: First submitted 2020-07-17; First posted 2020-08-18 (Actual); Results first posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Half of the participants will be randomized to receive the home-based PR with the mindful breathing module which consists of the Pursed Lipped Breathing Application and the Spire Health Tags (intervention) and half will receive the home-based PR (control).
Who Masked: Outcomes Assessor
Masking Description: Since the patients will know if they have the Pursed Lipped Breathing Application and Spire tags, the outcome assessor will be blinded to which arm received the Application and tags.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home-base pulmonary rehabilitation with mindful breathing modu (Experimental): Subjects will complete in a home-based pulmonary rehabilitation program and in addition will complete a mindful breathing practice using a module on a computer tablet.
  Interventions: Behavioral: Home-based pulmonary rehabilitation program; Behavioral: Mindful breathing module; Behavioral: Health coaching
- Home-base pulmonary rehabilitation (Active Comparator): Subjects will complete 12 week home-based pulmonary rehabilitation with health coaching
  Interventions: Behavioral: Home-based pulmonary rehabilitation program; Behavioral: Health coaching

INTERVENTIONS:
Behavioral: Home-based pulmonary rehabilitation program — Subjects will wear an activity monitor while doing at home exercises using a computer tablet
Behavioral: Mindful breathing module — Additional module on the computer tablet that involves inhaling and exhaling while following an animated ball on the computer screen.
  Arms: Home-base pulmonary rehabilitation with mindful breathing modu
Behavioral: Health coaching — Weekly coaching calls to discuss rehabilitation and health process using motivational interviewing

SUMMARY:
The purpose of this study is to develop a mindful breathing module to an already effective and developed home based rehabilitation program for guiding COPD patients in a mindful breathing practice and further palliate breathlessness and anxiety.

DETAILED DESCRIPTION:
A breathing technique called Pursed Lipped Breathing (PLB) has been proven to be beneficial for patients with COPD. PLB can ease shortness of breath and reduce stress and anxiety. This study will develop a mindful PLB module to compliment an already developed home based pulmonary rehabilitation program. In this study, patients will be randomized to either a group that does the home based pulmonary rehabilitation with the mindful breathing module and health coaching or a group that does the home based pulmonary rehabilitation with health coaching without the mindful breathing module. Both groups will do the home based pulmonary rehabilitation for 12 weeks. In addition there are questionnaires and the wearing of an activity monitor when you sign up and at 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Adults, age ≥ 40 years old.
* Clinical diagnosis of Chronic Obstructive Pulmonary Disease (COPD).
* At least 10 pack years of smoking.

Exclusion Criteria:

* Unable to do mild exercise (orthopedic-neurologic problems or confined to a bed).
* Unable to follow commands (cognitive impairment).
* Have a high likelihood of being lost to follow-up (active alcohol or drug abuse).
* Live in an area that does not have cellular service (Verizon).

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2021-08-06 (Actual); Primary Completion 2024-05-07 (Actual); Study Completion 2024-05-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roberto P Benzo, Principal Investigator — Mayo Clinic; Kevin Kramer, PhD, Principal Investigator — Minnesota HealthSolutions
Locations (2):
- United States (2):
  - Minnesota HealthSolutions Corporporation, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Home-base Pulmonary Rehabilitation With Mindful Breathing Module: Subjects completed a home-based pulmonary rehabilitation program and in addition completed a mindful breathing practice using a module on a computer tablet.
  Home-based pulmonary rehabilitation program: Subjects wore an activity monitor while doing at home exercises using a computer tablet
  Mindful breathing module: Additional module on the computer tablet that involved inhaling and exhaling while following an animated ball on the computer screen.
  Health coaching: Weekly coaching calls to discuss rehabilitation and health process using motivational interviewing
- Home-base Pulmonary Rehabilitation: Subjects completed a 12-week home-based pulmonary rehabilitation with health coaching
  Home-based pulmonary rehabilitation program: Subjects wore an activity monitor while doing at home exercises using a computer tablet
  Health coaching: Weekly coaching calls to discuss rehabilitation and health process using motivational interviewing
Period: Overall Study
Arm/Group | Home-base Pulmonary Rehabilitation With Mindful Breathing Module | Home-base Pulmonary Rehabilitation
Started | 48 | 51
Completed | 48 | 51
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Home-base Pulmonary Rehabilitation With Mindful Breathing Module | Home-base Pulmonary Rehabilitation | Total
Number analyzed (Participants) | 48 | 51 | 99
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.551 (6.894) | 70.103 (8.922) | 69.832 (7.957)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 29 | 58
  Male | 19 | 22 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 47 | 50 | 97
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 0 | 0 | 0
  White | 45 | 48 | 93
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 48 | 51 | 99

OUTCOME MEASURES:

1. Primary Outcome: Change in Chronic Respiratory Disease Questionnaire (CRQ)- Dyspnea Score
Description: The CRQ-Dyspnea is a 5-item questionnaire that assesses dyspnea on a Likert scale from 1 (Extremely short of breath) to 7 (Not at all short of breath). Total scores range from 5 - 35. Lower scores indicated higher severity of dyspnea. Higher scores indicate less severity of dyspnea.
Time Frame: Baseline, 3 months, 6 months
Population: For the Home-based pulmonary rehabilitation with mindful breathing module arm, nineteen subjects did not complete the three months or six months questionnaire. Data was not collected or analyzed.
  For the Home-base pulmonary rehabilitation arm, twenty-six subjects did not complete the three months questionnaire and twenty-eight subjects did not complete the six months questionnaire. Data was not collected or analyzed.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Home-base Pulmonary Rehabilitation With Mindful Breathing Module | Home-base Pulmonary Rehabilitation
Number analyzed (Participants) | 29 | 25
score on a scale
  baseline, 3 months | 0.68 [0.36 to 1.0] | 0.71 [0.19 to 1.22]
  baseline, 6 months: number analyzed (Participants) | 29 | 23
  baseline, 6 months | 0.34 [-0.03 to 0.71] | 0.83 [0.11 to 1.55]

2. Primary Outcome: Change in Chronic Respiratory Disease Questionnaire (CRQ)- Emotions Score
Description: The CRQ-Emotions is a 7-item questionnaire that assesses emotions on a Likert scale from 1 (All of the time) to 7 (None of the time). Total scores range from 7-49. Lower scores indicate more severity of emotions. Higher scores indicate less severity of emotions.
Time Frame: baseline, 3 months, 6 months
Population: For the Home-based pulmonary rehabilitation with mindful breathing module arm, nineteen subjects did not complete the three months or six months questionnaire. Data was not collected or analyzed.
  For the Home-base pulmonary rehabilitation arm, twenty-five subjects did not complete the three months questionnaire and twenty-eight subjects did not complete the six months questionnaire. Data was not collected or analyzed.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Home-base Pulmonary Rehabilitation With Mindful Breathing Module | Home-base Pulmonary Rehabilitation
Number analyzed (Participants) | 29 | 26
score on a scale
  baseline, 3 months | 0.45 [0.01 to 0.88] | 0.55 [0.14 to 0.97]
  baseline, 6 months | 0.35 [0.04 to 0.66] | 0.5 [-0.07 to 1.06]

3. Secondary Outcome: Change in Daily Physical Activity
Description: Mean change in the number of steps per day
Time Frame: baseline, 3 months, 6 months
Population: For the Home-based pulmonary rehabilitation with mindful breathing module arm, twenty-one subjects did not complete the three months or six months questionnaire. Data was not collected or analyzed.
  For the Home-base pulmonary rehabilitation arm, twenty-five subjects did not complete the three months questionnaire and thirty subjects did not complete the six months questionnaire. Data was not collected or analyzed.
Measure: Mean (95% Confidence Interval); unit: steps per day
Arm/Group | Home-base Pulmonary Rehabilitation With Mindful Breathing Module | Home-base Pulmonary Rehabilitation
Number analyzed (Participants) | 27 | 26
steps per day
  baseline, 3 months | 765.98 [46.16 to 1485.79] | 701.5 [-49.43 to 1452.43]
  baseline, 6 months: number analyzed (Participants) | 27 | 21
  baseline, 6 months | -181.78 [-987.65 to 624.09] | 290.36 [-537.44 to 1118.17]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline to end of study, approximately six months.
Arm/Group | Home-base Pulmonary Rehabilitation With Mindful Breathing Module | Home-base Pulmonary Rehabilitation
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/51
Other Adverse Events (participants affected / at risk) | 0/48 | 0/51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-08): https://cdn.clinicaltrials.gov/large-docs/00/NCT04517500/Prot_SAP_000.pdf